CLINICAL TRIAL: NCT01880996
Title: The Effect of Tai-chi/Qi-gong on Quality of Life (QOL), Sleep, and Fatigue in Patients With Gynecological Malignancies
Brief Title: Tai-chi / Qi-gong in Patients With Patients With Gynecological Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The deparment failed to detect patients that were willing to participate in this study
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dorit Gamus, Director, Complementary Medicine Service, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0112-DG-CTIL
Record Dates: First submitted 2013-05-30; First posted 2013-06-19 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Other Gynecological Cancers
Keywords: Ovarian Cancer; Gynecological Malignancies; Chemotherapy; Tai-chi; Qigong; Fatigue; Quality of life; Sleep disturbance
MeSH Terms: conditions — Ovarian Neoplasms; Fatigue; Parasomnias | interventions — Tai Ji; Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai-chi/Qi-gong (Experimental): 30 gynecological cancer patients scheduled for the first or second line of chemotherapy treatment will be recruited for this study to receive Tai-chi/qigong treatment initiated at the beginning of chemotherapy therapy, once a week (45 min each), for 10 weeks.
  Interventions: Other: Tai-chi/Qi-gong
- Usual Care (No Intervention): 30 gynecological cancer patients scheduled for primary or secondary chemotherapy treatment, will be evaluated by the same measures as the intervention group.

INTERVENTIONS:
Other: Tai-chi/Qi-gong — Tai-chi/Qi-gong employs a series of positions and movements that are performed in a slow, flowing manner to help a person concentrate on breathing and motion. The treatments will take place once a week at the Dept. of the Gyneco-oncology and the patients will be instructed to practice tai-chi at home on a daily basis
  Other Names: Tai Chi; Qi-gong; Taichi; Qigong
  Arms: Tai-chi/Qi-gong

SUMMARY:
Oncologic patients often report increased fatigue during and after chemotherapy. Evidence suggests Tai-chi/Qi-gong may improve quality of life (QOL) in oncologic patients treated with chemotherapy. Previous studies, mostly performed in a population of breast cancer patients, have demonstrated the benefits of Tai-chi/Qi-gong practice in improving quality of life (1), reducing bone resorption (2), preventing the decrease of blood counts (WBC and Hb) (3), and reducing inflammation (4).

The aim of this pilot study is to evaluate the effect of Tai-chi/Qi-gong on QOL, sleep, and fatigue in patients with gynecological malignancies, particularly in patients with ovarian cancer.

DETAILED DESCRIPTION:
Tai-chi/Qi-gong is a complementary medicine technique that synergizes the mind-body connection. The technique employs a series of positions and movements that are performed in a slow, flowing manner to help a person concentrate on breathing and motion.

The effect of Tai-chi/Qi-gong on fatigue, quality of life, and quality of sleep will be assessed in gynecological cancer patients. This trial will recruit 60 patients with gynecological malignancies, who receive first or second line chemotherapy. The patients will be allocated according to their preference to either the study or the control group. The Tai-chi/Qi-gong classes will take place once a week, for 10 consecutive weeks, at the facilities of the gyneco-oncology department. All patients will fill out the questionnaires at the beginning of the study, after 5 weeks, and upon the completion of the study (10 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Women with gynecological malignancies undergoing primary or secondary chemotherapy

Exclusion Criteria:

* Motor disability;
* Less than 1 month since the last abdominal surgery;
* Ascites

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in the Multidimensional Quality of Life Scale cancer MQOLS-CA | Week 0, Week 5, Week 10
  The Multidimensional Quality of Life Scale cancer MQOLS-CA was written by Padilla (5) and translated into Hebrew by Dorit Pud (6).

SECONDARY OUTCOMES:
Change in the Lee Fatigue Scale (LFS) | Week 0, Week 5, Week 10
  The Lee Fatigue Scale (LFS). The questionnaire was compiled by Lee (7) and translated into Hebrew by Dr. Dorit Pud (6).
Change in the Visual Analog Scale for Pain | Week 0, Week 5, Week 10

OTHER OUTCOMES:
Change in the White Blood Cell Count | Week 0, Week 3, Week 6, Week 9
  Results of the routine blood exams will be documented
Change in the Hemoglobin in blood | Week 0, Week 3, Week 6, Week 9
  Results of the routine blood exams will be documented
Change in the C-reactive protein in blood | Week 0, Week 3, Week 6, Week 9
Change in the Body Weight | Week 0, Week 5, Week 10
Change in the number of Emergency Room visits | Week 0, Week 5, Week 10
  Emergency Room visits for nausea, vomiting, or dehydration
Pattern of use of Complementary Medicine | Week 0, Week 5, Week 10
  List of Complementary modalities used including Medical Cannabis

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Gamus, M.D. Ph.D., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Hospital, Ramat Gan, Israel

REFERENCES:
- [Background] Oh B, Butow P, Mullan B, Clarke S, Beale P, Pavlakis N, Kothe E, Lam L, Rosenthal D. Impact of medical Qigong on quality of life, fatigue, mood and inflammation in cancer patients: a randomized controlled trial. Ann Oncol. 2010 Mar;21(3):608-614. doi: 10.1093/annonc/mdp479. Epub 2009 Oct 30. PMID 19880433
- [Background] Peppone LJ, Mustian KM, Janelsins MC, Palesh OG, Rosier RN, Piazza KM, Purnell JQ, Darling TV, Morrow GR. Effects of a structured weight-bearing exercise program on bone metabolism among breast cancer survivors: a feasibility trial. Clin Breast Cancer. 2010 Jun;10(3):224-9. doi: 10.3816/CBC.2010.n.030. PMID 20497921
- [Background] Yeh ML, Lee TI, Chen HH, Chao TY. The influences of Chan-Chuang qi-gong therapy on complete blood cell counts in breast cancer patients treated with chemotherapy. Cancer Nurs. 2006 Mar-Apr;29(2):149-55. doi: 10.1097/00002820-200603000-00012. PMID 16565626
- [Background] Padilla GV, Mishel MH, Grant MM. Uncertainty, appraisal and quality of life. Qual Life Res. 1992 Jun;1(3):155-65. doi: 10.1007/BF00635615. PMID 1301125
- [Background] Pud D, Ben Ami S, Cooper BA, Aouizerat BE, Cohen D, Radiano R, Naveh P, Nikkhou-Abeles R, Hagbi V, Kachta O, Yaffe A, Miaskowski C. The symptom experience of oncology outpatients has a different impact on quality-of-life outcomes. J Pain Symptom Manage. 2008 Feb;35(2):162-70. doi: 10.1016/j.jpainsymman.2007.03.010. Epub 2007 Dec 21. PMID 18082357
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970